CLINICAL TRIAL: NCT01987063
Title: National Prospective and Comparative Study on the Mode of Delivery of Twins
Acronym: JUMODA
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI12012
Record Dates: First submitted 2013-11-04; First posted 2013-11-19 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Pregnant Woman With Twins After 22 Weeks 0 Days of Gestation
Keywords: Twin delivery; Planned vaginal delivery; Planned cesarean delivery; Total breech extraction; Internal cephalic version; External cephalic version

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- pregnant woman with twins: pregnant woman with twins

SUMMARY:
The purpose of this study is to determine the best obstetrical practices for twin delivery.

DETAILED DESCRIPTION:
Large retrospective cohort studies have reported increased neonatal death and morbidity associated with vaginal delivery in comparison with cesarean in twin pregnancies. A recent large international randomized trial, the Twin Birth Study (TBS), showed that planned cesarean does not significantly decrease or increase the risk of fetal or neonatal death or serious neonatal morbidity, as compared with planned vaginal delivery in twin pregnancy between 32 and 39 weeks of gestation with a first twin in cephalic presentation. However, neither these large retrospective cohort studies, because information regarding delivery management is lacking, nor the TBS, because of insufficient statistical power, can answer the question on how to manage vaginal twin deliveries.

The aim of the JUMODA study is first to confirm in France whether planned vaginal delivery is not associated with increased neonatal risks in comparison with planned caesarean as shown in the TBS and secondly to determine the best obstetrical practices in case of vaginal delivery.

Analysis will be performed according to the planned mode of delivery (planned cesarean or planned vaginal delivery) and stratified according to:

1. Twin rank: second or first twin
2. Gestational age: before 28 weeks of gestation, before 32 weeks, after 32 weeks, and after 35 weeks
3. In the whole population and in low risk populations.

   For women delivering vaginally, analysis will be stratified according to:
4. Second twin presentation: vertex or non vertex
5. Obstetrical manoeuvres: none, internal cephalic version, external cephalic version, total breech extraction

ELIGIBILITY:
Inclusion Criteria:

* All patients delivering twins after 22 weeks and 0 days gestation in the participating maternities will be included in the study.

Exclusion Criteria:

* Patients who expressed opposition to the use of personal medical data or medical data from their children for this research will not be included in the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: cohort of pregnant woman with twins or triplets or quadruples
Sampling Method: Non-Probability Sample
Enrollment: 8979 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Composite measure of intrapartum and neonatal death and serious morbidity of the second twin after 32 weeks 0 days of gestation | 72 hours after birth
  * Intrapartum fetal death
  * Neonatal mortality
  * Apgar score lower than 4 at 5 minutes
  * Neonatal trauma (fracture of long bones or skull, subdural hematoma, brachial plexus elongation, phrenic or facial paralysis, injury of the spinal cord
  * Abnormal level of consciousness (coma, stupor, abnormal response to pain)
  * Intubation longer than 24 hours within the first 72 hours of life, two or more episodes of neonatal convulsions in the first 72 hours of life
  * Proved neonatal infection
  * Bronchopulmonary dysplasia
  * Necrotizing enterocolitis
  * Intraventricular hemorrhage grade III or IV
  * Periventricular leukomalacia.

SECONDARY OUTCOMES:
Composite measure of intrapartum and neonatal death and serious morbidity of the first twin after 32 weeks 0 days of gestation | Day 28 after birth
  Composite measure of intrapartum and neonatal death and serious morbidity of the first twin after 32 weeks 0 days of gestation
Composite measure of intrapartum and neonatal death and serious morbidity of the second twin after 32 weeks 0 days of gestation | Day 28 after birth
  Composite measure of intrapartum and neonatal death and serious morbidity of the second twin after 32 weeks 0 days of gestation
Composite measure of maternal death and serious morbidity after 32 weeks 0 days of gestation | Weeks after birth and before hospital discharge
  * Maternal death
  * Severe postpartum hemorrhage (PPH) defined as PPH requiring transfusion, embolisation, surgery, intensive care unit
  * Pulmonary embolism, deep venous thrombosis
  * Cerebrovascular accident
  * Postpartum psychosis
  * Severe thrombopenia (<50 000)
  * Severe anemia (<7g/dL)
  * Renal failure (oliguria <500 mL/24h or creatinin>135 mmol/L)
  * Maternal transfer in ICU
  * Laparotomy
  * Intraoperative injury to the bowel, ureter or bladder requiring repair
  * Vulvar or perineal hematoma requiring evacuation
  * Third and fourth degree perineal lacerations
  * Systemic infection (positive blood culture or temperature > 38.5 °C on two or more occasions at least 24h apart)
Duration of neonatal hospitalisation of first twin | Weeks after birth and before hospital discharge
  Duration between birth and hospital discharge
Duration of neonatal hospitalisation of second twin | Weeks after birth and before hospital discharge
  Duration between birth and hospital discharge
Duration of maternal hospitalisation | Weeks after birth and before hospital discharge
  Duration between delivery and hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: François GOFFINET, MD, PhD, Principal Investigator — APHP, France
Locations (1):
- Hôpital Robert Debré - APHP, Paris, France

REFERENCES:
- [Background] Barrett JF, Hannah ME, Hutton EK, Willan AR, Allen AC, Armson BA, Gafni A, Joseph KS, Mason D, Ohlsson A, Ross S, Sanchez JJ, Asztalos EV; Twin Birth Study Collaborative Group. A randomized trial of planned cesarean or vaginal delivery for twin pregnancy. N Engl J Med. 2013 Oct 3;369(14):1295-305. doi: 10.1056/NEJMoa1214939. PMID 24088091
- [Background] Smith GC. Perinatal death in twins. Author's reply on absolute risk. BMJ. 2007 Apr 14;334(7597):762. doi: 10.1136/bmj.39176.426424.3a. No abstract available. PMID 17436454
- [Background] Smith GC, Shah I, White IR, Pell JP, Dobbie R. Mode of delivery and the risk of delivery-related perinatal death among twins at term: a retrospective cohort study of 8073 births. BJOG. 2005 Aug;112(8):1139-44. doi: 10.1111/j.1471-0528.2005.00631.x. PMID 16045531
- [Background] Smith GC, Pell JP, Dobbie R. Birth order, gestational age, and risk of delivery related perinatal death in twins: retrospective cohort study. BMJ. 2002 Nov 2;325(7371):1004. doi: 10.1136/bmj.325.7371.1004. PMID 12411358
- [Result] Korb D, Schmitz T, Seco A, Goffinet F, Deneux-Tharaux C; JUmeaux MODe d'Accouchement (JUMODA) study group and the Groupe de Recherche en Obstetrique et Gynecologie (GROG). Risk factors and high-risk subgroups of severe acute maternal morbidity in twin pregnancy: A population-based study. PLoS One. 2020 Feb 28;15(2):e0229612. doi: 10.1371/journal.pone.0229612. eCollection 2020. PMID 32109258
- [Result] Korb D, Deneux-Tharaux C, Seco A, Goffinet F, Schmitz T; JUmeaux MODe d'Accouchement (JUMODA) study group and the Groupe de Recherche en Obstetrique et Gynecologie (GROG). Risk of Severe Acute Maternal Morbidity According to Planned Mode of Delivery in Twin Pregnancies. Obstet Gynecol. 2018 Sep;132(3):647-655. doi: 10.1097/AOG.0000000000002788. PMID 30095775
- [Result] Schmitz T, Prunet C, Azria E, Bohec C, Bongain A, Chabanier P, D'Ercole C, Deruelle P, De Tayrac R, Dreyfus M, Dupont C, Gondry J, Graesslin O, Kayem G, Langer B, Marpeau L, Morel O, Parant O, Perrotin F, Pierre F, Poulain P, Riethmuller D, Rozenberg P, Rudigoz RC, Sagot P, Senat MV, Sentilhes L, Vayssiere C, Venditelli F, Verspyck E, Winer N, Lecomte-Raclet L, Ancel PY, Goffinet F; JUmeaux MODe d'Accouchement (JUMODA) Study Group and the Groupe de Recherche en Obstetrique et Gynecologie (GROG). Association Between Planned Cesarean Delivery and Neonatal Mortality and Morbidity in Twin Pregnancies. Obstet Gynecol. 2017 Jun;129(6):986-995. doi: 10.1097/AOG.0000000000002048. PMID 28486364